CLINICAL TRIAL: NCT00141050
Title: Safety and Efficacy Study of Dexmethylphenidate in Children With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CRIT124EUS12
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: ADHD
Keywords: ADHD, children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dexmethylphenidate Hydrochloride

INTERVENTIONS:
Drug: Focalin XR

SUMMARY:
The purpose of this study is to compare the safety and efficacy of two doses of dexmethylphenidate to two doses of an approved, long-acting, marketed medication for ADHD (MPH) and placebo in children ages 6-12 diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of ADHD
* Males and females aged 6-12

Exclusion Criteria:

* Inability to understand or follow instructions
* Is pregnant
* Diagnosis of tic disorder
* History of seizure disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 2005-05; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change in attention and deportment measured at 2 hours post-dose

SECONDARY OUTCOMES:
Onset of effect at 0.5, 1, 2, 3, 4, 6, 8, 10, 11, and 12 hours post-dose
Parent's assessment of patient behavior across all treatment periods as measured by the change from baseline
Safety and tolerability of two doses of dexmethylphenidate compared to two doses of an approved, long-acting, marketed medication for ADHD and placebo in children ages 6-12 diagnosed with ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brams, MD, Principal Investigator — Bayou City Research
Locations (1):
- Bayou City Research, Houston, Texas, United States